CLINICAL TRIAL: NCT04015453
Title: Correlation of Early Postoperative Scar Appearance With Long-term Scar Outcomes: a Single Academic Institution Study
Brief Title: Correlation of Early Postoperative Scar Appearance With Long-term Scar Outcomes
Status: Completed | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 825545
Record Dates: First submitted 2019-07-09; First posted 2019-07-11 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Scar; Surgical Wound; Quality of Life; Mohs Micrographic Surgery; Skin Cancer Face
MeSH Terms: conditions — Cicatrix; Surgical Wound | interventions — Mohs Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Mohs micrographic surgery — All participants will have received Mohs micrographic surgical treatment for a facial skin cancer.

SUMMARY:
A retrospective cohort study of early and late period postoperative scars using previously validated survey measures and clinical photographs. The target population consists of participants treated with Mohs micrographic surgery (MMS) for a facial skin cancer by the division of dermatologic surgery. This study aims to determine if patient assessment of scar appearance correlates with physician ratings and/or third-person observer ratings. Secondary goals are to assess for correlations between early post-operative scar appearance and long-term scar appearance as well as identification of predictive factors for scar healing.

DETAILED DESCRIPTION:
Scarring is an inevitable outcome of surgical manipulation of the skin. Previous studies have shown that postoperative scarring, especially in cosmetically sensitive areas, may negatively affect patient quality of life and social interactions. The impact of surgical scarring is magnified in Mohs micrographic surgery, for which the large proportion of treated lesions are in highly visible areas, such as the head, face, and neck. Clinicians often underestimate the significance of scarring in patients' daily activities. Patients desire quick healing surgical scars in order to reintegrate into their normal social routines. Anecdotal evidence suggests that scars that heal well early in the post-operative period will achieve better results in the late postoperative period. Determining a model of early and late surgical scar evolution, as rated by patients, physicians, and third-party observers may; 1. Identify gaps between physician and patient evaluations; 2. Assist clinicians in effectively evaluating and counseling patients regarding their post-operative scar appearance.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants diagnosed with a biopsy-proven facial skin cancer (melanoma and non-melanoma skin cancers) and treated with Mohs micrographic surgery (MMS) from August 2015 to February 2016.

Exclusion Criteria:

* Participants with post-excisional reconstruction requiring multiple techniques, incomplete or missing patient photographs from postsurgical visits, or if the patient received any postoperative scar interventions (pulse-dye laser, scar revision, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult participants with a biopsy-proven facial skin cancer treated with MMS from 8/2015 to 2/2016.
Sampling Method: Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Physician Observer Scar Assessment Scale (POSAS) | 1 week postoperative measure
  The Patient and Observer Scar Assessment Scale (POSAS) is a validated scoring instrument that takes into account patient, physician, and third-party observer input to evaluate postsurgical scar quality in clinical photos. The instrument has 6 patient and 6 observer specific questions. Scoring of each question is performed on a scale of 1 to 10 where 1 is synonymous with "like normal skin" and 10 to the "worst scar imaginable". In addition, an overall total opinion score on a scale from 1 to 10 where 1 is akin to normal skin and 10 to the worst scar imaginable. Consequently, higher scores on either scale represent a worse scar appearance in the perception of the rater.
Physician Observer Scar Assessment Scale (POSAS) | 3 month postoperative measure
  Please refer to description above.

REFERENCES:
- [Background] Brown BC, McKenna SP, Siddhi K, McGrouther DA, Bayat A. The hidden cost of skin scars: quality of life after skin scarring. J Plast Reconstr Aesthet Surg. 2008 Sep;61(9):1049-58. doi: 10.1016/j.bjps.2008.03.020. Epub 2008 Jul 9. PMID 18617450
- [Background] Young VL, Hutchison J. Insights into patient and clinician concerns about scar appearance: semiquantitative structured surveys. Plast Reconstr Surg. 2009 Jul;124(1):256-265. doi: 10.1097/PRS.0b013e3181a80747. PMID 19568089
- [Background] Dey JK, Ishii LE, Byrne PJ, Boahene KD, Ishii M. The social penalty of facial lesions: new evidence supporting high-quality reconstruction. JAMA Facial Plast Surg. 2015 Mar-Apr;17(2):90-6. doi: 10.1001/jamafacial.2014.1131. PMID 25474194
- [Background] Draaijers LJ, Tempelman FR, Botman YA, Tuinebreijer WE, Middelkoop E, Kreis RW, van Zuijlen PP. The patient and observer scar assessment scale: a reliable and feasible tool for scar evaluation. Plast Reconstr Surg. 2004 Jun;113(7):1960-5; discussion 1966-7. doi: 10.1097/01.prs.0000122207.28773.56. PMID 15253184
- [Background] Shao K, Parker JC, Taylor L, Mitra N, Sobanko JF. Reliability of the Patient and Observer Scar Assessment Scale When Used With Postsurgical Scar Photographs. Dermatol Surg. 2018 Dec;44(12):1650-1652. doi: 10.1097/DSS.0000000000001479. No abstract available. PMID 29381545
- [Background] Sobanko JF, Zhang J, Margolis DJ, Etzkorn JR, Shin TM, Sarwer DB, Miller CJ. Patient-reported quality of life and psychosocial health prior to skin cancer treatment - A cross-sectional study. J Am Acad Dermatol. 2016 Jul;75(1):217-218.e2. doi: 10.1016/j.jaad.2016.01.033. No abstract available. PMID 27317520
- [Background] Zhang J, Miller CJ, O'Malley V, Bowman EB, Etzkorn JR, Shin TM, Sobanko JF. Patient and Physician Assessment of Surgical Scars: A Systematic Review. JAMA Facial Plast Surg. 2018 Jul 1;20(4):314-323. doi: 10.1001/jamafacial.2017.2314. PMID 29392275